CLINICAL TRIAL: NCT02619305
Title: Social Network Outcomes of a Livelihood Intervention for Impoverished Women in Rural Uganda: Randomized Controlled Trial
Brief Title: Social Network Outcomes of a Livelihood Intervention for Impoverished Women in Rural Uganda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MH096620-S5
Record Dates: First submitted 2015-08-15; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Indigency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (Experimental): Participants will be social network ties of women receiving a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises
  Interventions: Other: Social network tie
- Delayed treatment (No Intervention): Participants will be social network ties of women receiving no intervention but who will be placed on a waitlist to receive the intervention after a 12-month delay.

INTERVENTIONS:
Other: Social network tie — Participants will be social network ties of women receiving a livelihood intervention package consisting of a orientation and training and a loan package of chickens and associated implements to create poultry microenterprises.
  Arms: Immediate treatment

SUMMARY:
The objective of our study is to determine whether a livelihood intervention can change economic and psychosocial outcomes of social network ties and geographically proximate neighbors of impoverished women in rural Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility will be limited to all adults living in Nyakabare Parish (i.e., aged 18 years and older), including emancipated minors. Emancipated minors will be defined as persons living below 18 years of age who are married, are pregnant, live with a biological child in the household, or are responsible for their own livelihood.

Exclusion Criteria:

* Persons under the age of 18 (other than emancipated minors as described above) and persons who do not live within Nyakabare Parish will not be permitted to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Household Food Insecurity Access Scale | 12 months
  Scale items range from 0 (never) to 3 (more than 10 days in the past month)
Hopkins Symptom Checklist Scale | 12 months
  Scale items range from 1 (not at all) to 4 (very much)

SECONDARY OUTCOMES:
HIV Stigma Scale | 12 months
  Agreement (yes/no) with 15 statements about persons living with HIV (range, 0-15), to be assessed among social network ties of HIV-positive study participants
Norms about Intimate Partner Violence Scale | 12 months
  Agreement (yes/no) with 5 different statements about the acceptability of intimate partner violence under 5 different scenarios (range, 0-5)
Social Integration Scale | 12 months
  Frequency of participation in 11 different community groups: vocational, positive living, local council, water, village health, agricultural extension, savings, religious, women's, gardening (range, 0-11)
Social Capital Scale | 12 months
  Agreement (yes/no) with 4 questions about social trust and social cohesion (range, 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, PhD, Principal Investigator — Massachusetts General Hospital; Bernard Kakuhikire, MBA, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda